CLINICAL TRIAL: NCT04740307
Title: A Phase 2, Multicenter, Clinical Study to Evaluate the Safety and Efficacy of MK-1308A (Coformulated MK-1308/MK-3475) in Combination With Lenvatinib (E7080/MK-7902) in First-line Therapy of Participants With Advanced Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of Coformulated Pembrolizumab/Quavonlimab (MK-1308A) in Combination With Lenvatinib (E7080/MK-7902) in Advanced Hepatocellular Carcinoma (MK-1308A-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1308A-004; MK-1308A-004 (Other: MSD); jRCT2061210033 (Other: jRCT (Japan Registry of Clinical Trials)); 2023-505698-34-00 (Registry Identifier: EU CT); U1111-1292-3158 (Registry Identifier: UTN); 2020-004490-52 (EudraCT Number)
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: cytotoxic T-lymphocyte-associated protein 4 (CTLA-4); Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Death-Ligand 2 (PDL2, PD-L2); receptor tyrosine kinase inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab/Quavonlimab + Lenvatinib (Experimental): Participants receive pembrolizumab/quavonlimab via intravenous (IV) infusion every 6 weeks (Q6W) for up to 2 years, plus lenvatinib orally (based on actual body weight at screening) until progressive disease or unacceptable toxicity for up to 5 years. In the event of discontinuation of pembrolizumab/quavonlimab due to intolerable toxicity, re-initiation of treatment with pembrolizumab may be considered.
  Interventions: Biological: Pembrolizumab/Quavonlimab; Drug: Lenvatinib; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab/Quavonlimab — Pembrolizumab/Quavonlimab (400 mg/25 mg) administered via IV infusion Q6W.
  Other Names: MK-1308A
Drug: Lenvatinib — Lenvatinib 12 mg (body weight [BW] ≥60 kg) or 8 mg (BW <60 kg) administered orally every day (QD).
  Other Names: MK-7902
Biological: Pembrolizumab — Pembrolizumab (400 mg) administered via IV infusion Q6W, in the event of intolerable toxicity to pembrolizumab/quavonlimab.
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of fixed dose coformulated pembrolizumab/quavonlimab (MK-1308A) plus lenvatinib in a first line (1L) hepatocellular carcinoma (HCC) setting. No hypothesis testing will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Has an HCC diagnosis confirmed by radiology, histology, or cytology (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible)
* Has Barcelona Clinic Liver Cancer (BCLC) Stage C disease, or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach
* Has a Child-Pugh class A liver score within 7 days prior to first dose of study intervention.
* Has a predicted life expectancy of >3 months
* Has at least 1 measurable HCC lesion based on RECIST 1.1, confirmed by BICR
* Has an Eastern Cooperative Oncology Group Performance Score (ECOG PS) of 0 to 1 within 7 days prior to first dose of study intervention.
* Participants with controlled hepatitis B will be eligible as long as they meet the following criteria: antiviral therapy for Hepatitis B virus (HBV) must be given for at least 4 weeks and HBV viral load must be less than 500 IU/mL prior to first dose of study drug
* Has adequately controlled blood pressure with or without antihypertensive medications
* Has adequate organ function.

Exclusion Criteria:

* Has had esophageal or gastric variceal bleeding within the last 6 months.
* Has bleeding or thrombotic disorders or use of factor X inhibitors or anticoagulants requiring therapeutic international normalized ratio (INR) monitoring, e.g., warfarin or similar agents
* Has clinically apparent ascites on physical examination
* Has inferior vena cava or cardiac involvement of HCC based on imaging
* Has had clinically diagnosed hepatic encephalopathy in the last 6 months unresponsive to therapy
* Has medical contraindications that preclude all forms of contrast-enhanced imaging (computed tomography [CT] or magnetic resonance imaging [MRI])
* Has gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib
* Has a preexisting Grade ≥3 gastrointestinal or non-gastrointestinal fistula
* Has clinically active hemoptysis (bright red blood of a least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug
* Has clinically significant cardiovascular impairment within 12 months of the first dose of study intervention, including New York Heart Association (NYHA) Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability
* Has had major surgery to the liver within 4 weeks prior to the first dose of study intervention
* Has had a minor surgery (i.e., simple excision) within 7 days prior to the first dose of study intervention (Cycle 1 Day 1)
* Has serious nonhealing wound, ulcer, or bone fracture
* Has received any systemic chemotherapy, including anti- vascular endothelial growth factor (VEGF) therapy, or any systemic investigational anticancer agents for treatment of HCC
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Has received locoregional therapy to liver within 4 weeks prior to the first dose of study intervention
* Has received prior radiotherapy to a non-liver region within 2 weeks of start of study intervention
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study drug
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has a known history of, or any evidence of, central nervous system (CNS) metastases and/or carcinomatous meningitis as assessed by local site investigator
* Has severe hypersensitivity (≥Grade 3) to study intervention and/or any of their excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy, with the exception of HBV or Hepatitis C virus (HCV)
* Has a known history of human immunodeficiency virus (HIV) infection
* Has dual active HBV infection (HBsAg (+) and /or detectable HBV DNA) and HCV infection (anti-HCV antibody [Ab] positive and detectable HCV RNA) at study entry
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with the participants ability to cooperate with the requirements of the study
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with a Dose-Limiting Toxicity (DLT) in the Safety Lead-in Phase | Cycle 1 (Up to approximately 3 weeks)
  DLTs will be defined as follows unless determined to be unrelated to study intervention: any Grade 4 nonhematologic toxicity (not laboratory); any Grade 4 hematologic toxicity lasting >7 days (Grade 4 lymphopenia lasting ≥21 days); Grade 3 platelet count decreased if associated with clinically significant hemorrhage; any Grade 3 nonhematologic toxicity (not laboratory) lasting >3 days despite optimal supportive care; any clinically significant Grade 3 or Grade 4 nonhematologic laboratory abnormality if: medical intervention is required to treat participant, or abnormality leads to hospitalization, or abnormality persists for >1 week (or bilirubin if persists >4 weeks); aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) >10.0 times upper limit of normal (ULN) or >10.0 times baseline if baseline >ULN; any febrile neutropenia Grade 3 or Grade 4; any treatment-related AE that causes the participant to discontinue study intervention during the DLT window; any Grade 5 toxicity
Number of participants with ≥1 adverse event (AE) | Up to approximately 5 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants with an AE will be reported.
Number of participants with ≥1 serious adverse event (SAE) | Up to approximately 5 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event. The number of participants with an SAE will be reported.
Number of participants with ≥1 immune-related AE (irAE) | Up to approximately 5 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. AEs associated with MK-1308A exposure may represent an immune-related response. irAEs pre-specified for this study include pneumonitis, diarrhea/colitis, Type 1 diabetes mellitus (T1DM) or hyperglycemia, hypophysitis, hyperthyroidism, hypothyroidism, nephritis (grading according to increased creatinine or acute kidney injury), and myocarditis. The number of participants with an irAE will be reported.
Number of participants with ≥1 hepatic AE | Up to approximately 5 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Hepatic events of clinical interest (ECIs) include any of the following events if the event is considered not due to disease progression as judged by the investigator: among participants with Baseline ALT <2 × ULN: ALT ≥5 × ULN; among participants with Baseline ALT ≥2 × ULN: ALT >3 × the Baseline level; ALT >500 U/L regardless of baseline level; total bilirubin >3.0 mg/dL; hepatic decompensation diagnosed clinically (regardless of laboratory values) including new onset clinically detectable ascites requiring intervention for >3 days, hepatic encephalopathy, or gastrointestinal bleeding suggestive of portal hypertension. The number of participants with a hepatic AE will be reported.
Number of participants discontinuing study treatment due to an AE | Up to approximately 5 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants that discontinue study treatment due to an AE will be reported.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR) | Up to approximately 28 months
  ORR is defined as the percentage of participants who achieve a confirmed Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters [SOD] of target lesions) per RECIST 1.1 adjusted for this study to allow a maximum of 10 target lesions in total and 5 per organ, and assessed by BICR.

SECONDARY OUTCOMES:
Duration of Response (DOR) per RECIST 1.1 as assessed by BICR | Up to approximately 28 months
  For participants who demonstrate confirmed CR or PR per RECIST 1.1 assessed by BICR, DOR is defined as the time from the first documented evidence of CR (disappearance of all target lesions) or PR (at least a 30% decrease in the SOD of target lesions) until progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1 adjusted for this study to allow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as at least a 20% increase in the SOD of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
Disease Control Rate (DCR) per RECIST 1.1 as assessed by BICR | Up to approximately 28 months
  DCR is defined as the percentage of participants who have achieved CR (disappearance of all target lesions), PR (at least a 30% decrease in the SOD of target lesions), or stable disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD) after ≥6 weeks (the start of the window for the first scheduled scan) per RECIST 1.1 assessed by BICR. Per RECIST 1.1 adjusted for this study to allow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as at least a 20% increase in the SOD of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
Progression Free Survival (PFS) per RECIST 1.1 as assessed by BICR | Up to approximately 28 months
  PFS is defined as the time from the first dose of study intervention to the first documented PD per RECIST 1.1 by BICR or death due to any cause, whichever occurs first. Per RECIST 1.1 adjusted for this study to allow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as at least a 20% increase in the SOD of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
Time-To-Progression (TTP) per RECIST 1.1 as assessed by BICR | Up to approximately 28 months
  TTP is defined as the time from the first dose of study intervention to the first documented PD per RECIST 1.1 assessed by BICR. Per RECIST 1.1 adjusted for this study to allow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as at least a 20% increase in the SOD of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
Overall Survival (OS) | Up to approximately 28 months
  OS is defined as the time from the first dose of study intervention to death due to any cause.
ORR per modified RECIST (mRECIST) as assessed by BICR | Up to approximately 28 months
  ORR is defined as the percentage of participants who achieve a confirmed CR (disappearance of any intratumoral arterial enhancement in all target lesions) or a PR (at least a 30% decrease in the SOD of viable [contrast enhancement in the arterial phase] target lesions, taking as reference the baseline SOD of target lesions) per mRECIST as assessed by BICR. mRECIST for HCC allows evaluation of treatment effects that are not reflected in simple total size changes of lesions.
DOR per mRECIST as assessed by BICR | Up to approximately 28 months
  For participants who demonstrate confirmed CR or PR per mRECIST assessed by BICR, DOR is defined as the time from the first documented evidence of CR (disappearance of any intratumoral arterial enhancement in all target lesions) or PR (at least a 30% decrease in the SOD of viable [contrast enhancement in the arterial phase] target lesions, taking as reference the baseline SOD of target lesions) until PD or death due to any cause, whichever occurs first. mRECIST for HCC allows evaluation of treatment effects that are not reflected in simple total size changes of lesions. Per mRECIST, PD was defined as an increase of at least 20% in the SODs of viable (enhancing) target lesions, taking as reference the smallest SODs of viable (enhancing) target lesions recorded since the treatment started.
DCR per mRECIST as assessed by BICR | Up to approximately 28 months
  DCR is defined as the percentage of participants who have achieved CR (disappearance of any intratumoral arterial enhancement in all target lesions), PR (at least a 30% decrease in the SOD of viable [contrast enhancement in the arterial phase] target lesions, taking as reference the baseline SOD of target lesions), or SD (any cases that do not qualify for either PR or PD) after ≥6 weeks (the start of the window for the first scheduled scan) per mRECIST assessed by BICR. mRECIST for HCC allows evaluation of treatment effects that are not reflected in simple total size changes of lesions. Per mRECIST, PD was defined as an increase of at least 20% in the SODs of viable (enhancing) target lesions, taking as reference the smallest SODs of viable (enhancing) target lesions recorded since the treatment started.
PFS per mRECIST as assessed by BICR | Up to approximately 28 months
  PFS is defined as the time from the first dose of study intervention to the first documented PD per mRECIST by BICR or death due to any cause, whichever occurs first. mRECIST for HCC allows evaluation of treatment effects that are not reflected in simple total size changes of lesions. Per mRECIST, PD was defined as an increase of at least 20% in the SODs of viable (enhancing) target lesions, taking as reference the smallest SODs of viable (enhancing) target lesions recorded since the treatment started.
TTP per mRECIST as assessed by BICR | Up to approximately 28 months
  TTP is defined as the time from the first dose of study intervention to the first documented PD per mRECIST assessed by BICR. mRECIST for HCC allows evaluation of treatment effects that are not reflected in simple total size changes of lesions. Per mRECIST, PD was defined as an increase of at least 20% in the SODs of viable (enhancing) target lesions, taking as reference the smallest SODs of viable (enhancing) target lesions recorded since the treatment started.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (40):
- United States (7):
  - City of Hope Comprehensive Cancer Center ( Site 0002), Duarte, California
  - Johns Hopkins Hospital-Sidney Kimmel Comprehensive Cancer Center - GI and Immunology ( Site 0013), Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai ( Site 0009), New York, New York
  - Oregon Health and Science University ( Site 0006), Portland, Oregon
  - Charleston Oncology ( Site 0003), Charleston, South Carolina
  - Blue Ridge Cancer Care ( Site 0008), Roanoke, Virginia
  - Virginia Mason Medical Center ( Site 0004), Seattle, Washington
- China (9):
  - Anhui Provincial Hospital ( Site 0113), Hefei, Anhui
  - Beijing Cancer hospital-Department of Hepato-Pancreato-Biliary Surgery II ( Site 0107), Beijing, Beijing Municipality
  - Fuzhou General hospital of Nanjing Military Command-Oncology Department ( Site 0105), Fuzhou, Fujian
  - Southern Medical University Nanfang Hospital-Liver Cancer Department ( Site 0106), Guangzhou, Guangdong
  - Wuhan Union Hospital Cancer Center ( Site 0108), Wuhan, Hubei
  - Hunan Cancer Hospital-intervention department ( Site 0109), Changsha, Hunan
  - The First Affiliated Hospital of Xian Jiaotong University ward1 depattment of medical oncology ( Sit, Xi'an, Shaanxi
  - Zhongshan Hospital,Fudan University ( Site 0103), Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated Fudan University-Surgery Department ( Site 0118), Shanghai, Shanghai Municipality
- Italy (3):
  - Humanitas-U.O di Oncologia medica ed Ematologia ( Site 0231), Rozzano, Milano
  - Ospedale San Raffaele-Oncologia Medica ( Site 0227), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-Department of Abdominal Oncology ( Site 0230), Napoli
- Japan (4):
  - National Cancer Center Hospital East ( Site 0153), Kashiwa, Chiba
  - Toranomon Hospital Kajigaya ( Site 0154), Kawasaki, Kanagawa
  - Kindai University Hospital- Osakasayama Campus-Department of Gastroenterology and Hepatology ( Site, Sayama, Osaka
  - Hiroshima University Hospital ( Site 0156), Hiroshima
- Poland (4):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Onkologii i Radioterapii ( Site, Warsaw, Masovian Voivodeship
  - Wojewódzki Szpital im. Św. Ojca Pio w Przemyślu ( Site 0249), Przemyśl, Podkarpackie Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 0247), Gdansk, Pomeranian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 0246), Koszalin, West Pomeranian Voivodeship
- South Korea (3):
  - Seoul National University Bundang Hospital-Medical Oncology ( Site 0290), Seongnam, Kyonggi-do
  - Samsung Medical Center ( Site 0288), Seoul, Kyonggi-do
  - Asan Medical Center ( Site 0289), Seoul
- Spain (2):
  - Hospital Universitario Central de Asturias-Hepatology ( Site 0309), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron-Liver Unit - Department of Internal Medicine ( Site 0310), Barcelona
- Switzerland (5):
  - Hôpitaux Universitaires de Genève (HUG) ( Site 0335), Geneva, Canton of Geneva
  - Cantonal Hospital St.Gallen-Klinik für Gastroenterologie / Hepatologie ( Site 0334), Sankt Gallen, Canton of St. Gallen
  - CHUV (centre hospitalier universitaire vaudois) ( Site 0333), Lausanne, Canton of Vaud
  - UniversitätsSpital Zürich-Gastroenterologie & Hepatologie ( Site 0332), Zurich, Canton of Zurich
  - Inselspital Bern-Universitätsklinik für Viszerale Chirurgie und Medizin ( Site 0331), Bern
- Taiwan (3):
  - NATIONAL CHENG-KUNG UNI. HOSP.-Clinical Trial Research Team of Liver Diseases ( Site 0354), Tainan
  - National Taiwan University Hospital-Oncology ( Site 0351), Taipei
  - Taipei Veterans General Hospital-Division of Gastroenterology & Hepatology, Department of Medicine (, Taipei

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com